CLINICAL TRIAL: NCT06519409
Title: Comparative Treatment Evaluation of Human Mandibular Class II Furcation Defects Using Bone Grafts and Antimicrobial Photodynamic Therapy-A Randomized Control Trial.
Brief Title: Comparison of Bone Graft and Photodynamic Therapy in Class II Furcation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCDS/185/PG/2015-16
Record Dates: First submitted 2023-07-26; First posted 2024-07-25 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Furcation Defects
MeSH Terms: conditions — Furcation Defects | interventions — Photochemotherapy

ARMS (1):
- Photodynamic therapy (Experimental): After debridement photodynamic therapy was performed by applying indocyanine green photo sensitizer to furcation defect sites for 1 min. A diode laser with the wavelength of 810 nm and 100 mW 0f power output in the continuous mode was applied to this site. The indocyanine dye has high absorption in the infrared spectrum with an absorption peak near 810 nm, which is close to the emission of diode lasers. This dye has low toxicity, a rapid elimination time and is a good photo sensitizer. The furcation defects then received the graft hydrated with sterile saline. The graft material compacted into the bone defect was similar to the control site.
  Interventions: Procedure: Open flap debridement and photodynamic therapy

INTERVENTIONS:
Procedure: Open flap debridement and photodynamic therapy

SUMMARY:
This is a surgical comparative clinical trial which aims to assess class II buccal furcation defects treated with Xenograft alone or preceded by antimicrobial photodynamic therapy.

DETAILED DESCRIPTION:
To test the efficacy of photodynamic therapy (Indocyanine green) along with placement of xenograft (Cerabone®-Natural bovine bone grafting material, Botiss biomaterials) to treat a class II furcation defects. The topical study was designed as a randomized controlled, single blinded (patient), split mouth clinical trial with 14 participants. In the control group, the defects were filled with xenograft (Cerabone®) whereas the test group received photodynamic therapy (Indocyanine green) in addition to grafting. Radiovisiography technique was used to observe the possible changes in the furcation region at baseline and 9 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy subjects Age group of 25-60 years Presence of class II furcation defect on buccal surfaces of mandibular molars as determined by clinical and radiographic evaluation.

Vertical probing depth (VPD) ≥4mm Horizontal probing depth (HPD) ≥4 mm Gingival margin (GM) coronal to or at the level of the roof of the furcation

Exclusion Criteria:

Current and former smokers Administration of antibiotics in the last 6 months History of any periodontal therapy in the past 6 months Known allergic responses to bovine derived graft materials and photosensitizers.

Pregnant and lactating women.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04-08 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
percentage of bone fill | 9 months
  amount of bone formation

SECONDARY OUTCOMES:
Clinical efficacy | 9 months
  clinical attachment level

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Prabhuji MLV, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: No